CLINICAL TRIAL: NCT01684436
Title: Safety and Efficacy of Punctal Plug Insertion in Patients With Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APMA-DE-0812
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Punctal Plugs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Punctal plug (Experimental): Punctal plugs inserted into the study eye on Day 1.
  Interventions: Device: Punctal Plug

INTERVENTIONS:
Device: Punctal Plug — Punctal plugs inserted into the study eye on Day 1.

SUMMARY:
This study will access changes in tear protein levels and symptoms of dry eye following insertion of a punctal plug.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe dry eye

Exclusion Criteria:

* Previous punctal plug insertion in the last 3 months or presence of plugs at the time of study
* Contact lens wear in the 7 days prior to study start or during the study
* LASIK procedure in the last year
* Cataract or other eye surgery in the last 3 months
* Corneal grafts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2013-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Singapore, Singapore

REFERENCES:
- [Background] Tong L, Beuerman R, Simonyi S, Hollander DA, Stern ME. Effects of Punctal Occlusion on Clinical Signs and Symptoms and on Tear Cytokine Levels in Patients with Dry Eye. Ocul Surf. 2016 Apr;14(2):233-41. doi: 10.1016/j.jtos.2015.12.004. Epub 2016 Jan 13. PMID 26774908

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Punctal Plug
Started | 30
Completed | 29
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: The number of participants for analysis includes all patients who completed the study
Arm/Group | Punctal Plug
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Tear Cytokine Levels Before Punctal Plug Insertion in the Study Eye
Description: A punctal plug (tear duct plug) is a device inserted into the tear duct (puncta) of the eye to block the tear duct from draining liquid from the eye. Tears were collected using the Schirmer's test strip. Tears are measured in the study eye for tear cytokine levels before punctal plug insertion in picogram(pg)/milliliter (mL)/millimeter (mm) of Schirmer's test strip moistened. Cytokines help with the generation of an immune response. Increased cytokine levels are representative of inflammation in the eye.
Time Frame: Week 0 (Baseline)
Population: All patients who completed the study
Measure: Mean (Standard Deviation); unit: picogram/milliliter/millimeter(pg/ml/mm)
Arm/Group | Punctal Plug
Number analyzed (Participants) | 29
picogram/milliliter/millimeter(pg/ml/mm)
  Interferon (IFN) | 2.24 (2.02)
  Interleukin-10 (IL10) | 4.69 (3.54)
  Interleukin-12 (IL12) | 9.08 (9.98)
  Interleukin-13 (IL13) | 29.81 (26.53)
  Interleukin-17A (IL17A) | 0.57 (0.48)
  Interleukin-1B (IL1B) | 0.63 (0.37)
  Matrix metallopeptidase 9 (MMP9) | 1519.82 (1516.92)
  Interleukin-2 (IL2) | 0.88 (0.59)
  Interleukin-4 (IL4) | 17.66 (21.59)
  Interleukin-6 (IL6) | 6.11 (6.73)
  Interleukin-8 (IL8) | 74.00 (55.03)
  Interferon γ-Induced Protein-10 (IP10) | 2384.86 (1198.08)
  Monocyte Chemotactic Protein 1 (MCP1) | 49.08 (46.91)
  Macrophage Inflammatory Protein 1 Alpha (MIP1A) | 0.59 (0.56)
  Regulate Activation Normal T-Cell Express (RANTE) | 21.20 (15.57)
  Tumor Necrosis Factor Alpha (TNFA) | 1.54 (1.46)

2. Secondary Outcome: Corneal Fluorescein Staining Score in the Study Eye
Description: The cornea is evaluated following ocular administration of fluorescein stain in the study eye. The cornea is the transparent front part of the eye which covers the iris and pupil. The cornea is divided into 5 regions. Each region is scored according to the extent of staining, with scores ranging from 0 to 4 points: 0=non-staining to 4=regional whole staining of the cornea with 0.5 unit intervals. The higher the staining score, the worse the dry eye condition.
Time Frame: Week 0 (Baseline), Week 3
Population: All patients who completed the study
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Punctal Plug
Number analyzed (Participants) | 29
Scores on a Scale
  Week 0 (Baseline): Superior | 0.57 (0.85)
  Week 0 (Baseline): Inferior | 1.33 (0.93)
  Week 0 (Baseline): Nasal | 0.67 (0.89)
  Week 0 (Baseline): Temporal | 0.72 (0.96)
  Week 0 (Baseline): Central | 0.91 (0.95)
  Week 3: Superior | 0.48 (0.62)
  Week 3: Inferior | 1.22 (0.85)
  Week 3: Nasal | 0.41 (0.84)
  Week 3: Temporal | 0.36 (0.74)
  Week 3: Central | 0.57 (0.73)

3. Secondary Outcome: Tear Film Break-up Time (TBUT)
Description: TBUT is defined as the time to initial breakup of the tear film following a blink. The longer it takes, the more stable the tear film.
Time Frame: Week 0 (Baseline), Week 3
Population: All patients who completed the study
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Punctal Plug
Number analyzed (Participants) | 29
Seconds
  Week 0 (Baseline) | 2.21 (0.57)
  Week 3 | 2.42 (0.76)

4. Secondary Outcome: Schirmer's Test Score
Description: The Schirmer's Test measures the rate of tear secretion by the eye over 5 minutes (min). The results indicate the presence of dry eye (Normal = greater than or equal to 10 millimeters (mm) of tears, Dry Eye = less than 10 mm of tears). The smaller the number, the more severe the dry eye.
Time Frame: Week 0 (Baseline), Week 3
Population: All patients who completed the study
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Punctal Plug
Number analyzed (Participants) | 29
Millimeters (mm)
  Week 0 (Baseline) | 5.07 (2.76)
  Week 3 | 6.28 (5.11)

5. Secondary Outcome: Dry Eye Questionnaire Irritation Score
Description: Severity of dry eye irritation is rated by the patient using a visual analogue scale (VAS). Patients put a mark on a 100 millimeter line where 0 (far left on the line)=no symptoms to 100 (far right on the line)=most severe symptoms. The higher the score, the more severe the symptoms.
Time Frame: Week 0 (Baseline), Week 3
Population: All patients who completed the study
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Punctal Plug
Number analyzed (Participants) | 29
Millimeters (mm)
  Week 0 (Baseline) | 53.81 (26.5)
  Week 3 | 36.22 (24.89)

6. Primary Outcome: Concentration of Tear Cytokine Levels Following Punctal Plug Insertion in the Study Eye
Description: as for outcome 1
Time Frame: Week 3
Population: All patients who completed the study
Measure: Mean (Standard Deviation); unit: picogram/milliliter/millimeter(pg/ml/mm)
Arm/Group | Punctal Plug
Number analyzed (Participants) | 29
picogram/milliliter/millimeter(pg/ml/mm)
  IFN | 3.12 (2.69)
  IL10 | 3.97 (3.35)
  IL12 | 7.34 (6.05)
  IL13 | 29.14 (23.35)
  IL17A | 0.55 (0.39)
  IL1B | 1.10 (1.03)
  MMP9 | 1445.53 (1415.09)
  IL2 | 1.05 (1.10)
  IL4 | 9.75 (8.31)
  IL6 | 4.31 (3.66)
  IL8 | 61.07 (57.15)
  IP10 | 2769.17 (1479.50)
  MCP1 | 68.08 (62.10)
  MIP1A | 0.61 (0.73)
  RANTE | 29.55 (26.99)
  TNFA | 1.37 (1.21)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected over the 3 week study period.
Description: All patients enrolled in the study were used for the analysis of adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | Punctal Plug
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.